CLINICAL TRIAL: NCT01691638
Title: Genetics of Periodontal Diseases in European Caucasians
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Kiel (Other)
Collaborators: Interleukin Genetics, Inc. (Industry)
Other Study IDs: ILI-11-127-PST2Europe
Record Dates: First submitted 2012-09-24; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Periodontitis
- Control

SUMMARY:
(A retrospective case control study to validate the association between Interleukin-1 gene variations and adult chronic periodontal disease in European Caucasians)

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: Dutch or German Caucasian

Exclusion Criteria:

* None (however, diabetics were excluded during original patient recruitment at several clinical sites).

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All study subjects will be selected from pre-existing patient databases in Germany and the Netherlands. All chronic periodontitis cases and controls will be subjects who were at least 35 years old at time of enrollment. Classification of chronic periodontitis will be based on extent of alveolar bone loss with consideration of tooth loss.
Sampling Method: Non-Probability Sample